CLINICAL TRIAL: NCT00403390
Title: Generic vs. Name-Brand Levothyroxine: Assessment of Bioequivalence Using TSH as a Marker in Children With Permanent Hypothyroidism
Brief Title: Generic vs. Name-Brand Levothyroxine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jeremi Carswell, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-11-146
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Congenital Hypothyroidism; Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brand name levothyroxine (Synthroid) (Experimental): Dose previously demonstrated to normalize thyroid function given daily for 2 months
  Interventions: Drug: Brand Name Levothyroxine (Synthroid)
- Generic formulation of Levothyroxine (Active Comparator): Dosage previously determined to normalize thyroid function given daily for 2 months
  Interventions: Drug: Generic formulation of Levothyroxine

INTERVENTIONS:
Drug: Brand Name Levothyroxine (Synthroid) — Randomized crossover study using 8 weeks of brand name levothyroxine (Synthroid, manufactured by Abbott), then 8 weeks of the generic formulation of levothyroxine (manufactured by Sandoz). The dose of medication does not change throughout the duration of the study.
  Other Names: Levothyroxine
  Arms: Brand name levothyroxine (Synthroid)
Drug: Generic formulation of Levothyroxine — Randomized crossover study using 8 weeks of the generic formulation of levothyroxine (manufactured by Abbott, then 8 weeks of brand name levothyroxine (Synthroid, manufactured by Abbott). The dose of medication does not change throughout the duration of the study.
  Other Names: No other names
  Arms: Generic formulation of Levothyroxine

SUMMARY:
This study compares two different brands of thyroxine (thyroid hormone). Currently, pharmacists may be substituting generic formulations of thyroid hormone without your doctor knowing about this. Although a small difference in thyroid function is not significant in most healthy children, adolescents and adults, in infants and toddlers even a small difference in thyroid function can have important harmful consequences on brain development. The purpose of the present study is to learn whether the difference between brands of thyroid hormone that are currently being substituted is sufficient to cause a difference in thyroid function.

DETAILED DESCRIPTION:
This study is an unblinded, randomized controlled cross-over study, which involves taking 2 different forms of levothyroxine sequentially over a 16 week period. Subjects will have a total of 3 visits over this time period. At the first visit, subjects are randomized to receive either generic (Sandoz) levothyroxine or Synthroid (Abbott) brand of levothyroxine. Blood is drawn for baseline thyroid function studies and other markers which are influenced by thyroid hormone at each visit. The second visit is the cross-over visit, and the final visit is a close-out visit, after which each subject will resume taking their previous formulation of levothyroxine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 18 years
* Diagnosis of Congenital Hypothyroidism with initial TSH > 100
* Ability to understand directions and follow all instructions

Exclusion Criteria:

* Not on any drug interfering with absorption of levothyroxine

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind S Brown, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Nothing currently planned

REFERENCES:
- [Result] Carswell JM, Gordon JH, Popovsky E, Hale A, Brown RS. Generic and brand-name L-thyroxine are not bioequivalent for children with severe congenital hypothyroidism. J Clin Endocrinol Metab. 2013 Feb;98(2):610-7. doi: 10.1210/jc.2012-3125. Epub 2012 Dec 21. PMID 23264396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through flyers in the endocrine clinic and letters with opt-out cards to contact. Recruitment started November 2006 and completed ended March 2010.
Pre-assignment Details: Subjects' ages had to be between 3-18 years and had a diagnosis of hypothyroidism, either congenital or acquired with an initial TSH of >100 uIU/mL.
Groups:
- Group 1: Branded Synthroid 8 weeks, then generic levothyroxine 8 weeks
- Group 2: Generic levothyroxine for 8 weeks then branded Synthroid for 8 weeks
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 16 | 18
Completed | 13 | 18
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — samples lost | 1 | 0
Not completed — non-compliant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Generic levothyroxine 8 weeks, then branded Synthroid 8 weeks
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 13 | 18 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 18 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (1.2) | 10 (1.0) | 10 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Thyroid Stimulating Hormone as Primary Endpoint Measured at Initiation of Study, After 8 Weeks of One Drug, and Then 8 Weeks After the Second Drug.
Time Frame: 3 points over 16 weeks
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 13 | 18
uIU/mL
  Baseline | 2.455 (1.532) | 2.131 (1.322)
  After first drug | 0.788 (0.631) | 3.053 (1.233)
  After second drug | 3.112 (4.983) | 1.217 (2.832)

ADVERSE EVENTS:
Groups:
- Group 1: Crossover; Branded Synthroid 8 weeks, then generic levothyroxine 8 weeks
- Group 2: Crossover; Generic levothyroxine 8 weeks, then Branded Synthroid 8 weeks, then generic
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18
Other Adverse Events (participants affected / at risk) | 0/13 | 0/18

LIMITATIONS AND CAVEATS:
Proof of principle study; small sample. Results may not be applicable to all populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes